CLINICAL TRIAL: NCT04576013
Title: Peripheral Nerve Stimulation to Improve Upper Extremity Function After Severe Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving the university.
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Lumy Sawaki, Associate Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 44185
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: neuroplasticity; rehabilitation; peripheral nerve stimulation; motor training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active PNS during training (Experimental): Individuals in this group will receive active PNS while participating in 2 hours of motor training of the affected arm.
  Interventions: Device: Peripheral nerve stimulation (PNS); Behavioral: Intensive upper extremity motor training
- Active PNS before training (Active Comparator): Individuals in this group will receive 2 hours of active PNS before participating in 2 hours of motor training of the affected arm.
  Interventions: Device: Peripheral nerve stimulation (PNS); Behavioral: Intensive upper extremity motor training
- Sham PNS during training (Sham Comparator): Individuals in this group will receive 2 hours of sham PNS while participating in 2 hours of motor training of the affected arm.
  Interventions: Device: Peripheral nerve stimulation (PNS); Behavioral: Intensive upper extremity motor training

INTERVENTIONS:
Device: Peripheral nerve stimulation (PNS) — Non-invasive stimulation is applied to 3 nerves of the arm. The stimulation will be set at a level that is not painful or uncomfortable.
Behavioral: Intensive upper extremity motor training

SUMMARY:
Subjects will receive non-invasive stimulation of nerves on their arm and intensive motor training of their arm. The timing of the stimulation in relation to the training will vary by group.

DETAILED DESCRIPTION:
This study will look at the differences in improvement of hand and arm function when nerve stimulation is applied at different times in relation to motor training. The nerve stimulation, called peripheral nerve stimulation (PNS), is non-invasive and painless. Subjects in the study may receive strong or mild PNS. Subjects will also vary by whether PNS is delivered for 2 hours before the 2 hours of motor training, or during the 2 hours of motor training. Which level of stimulation and its timing will be determined randomly for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Have severe upper extremity motor deficit after a single stroke
* Stroke onset at least 12 months ago

Exclusion Criteria:

* Addition or change in the dosage of drugs known to exert detrimental effects on motor recovery within 3 months of enrollment
* Untreated depression
* History of multiple strokes
* History of seizure
* History of head injury with loss of consciousness, severe alcohol or drug abuse, or psychiatric illness
* Positive pregnancy test or being of childbearing age and not using appropriate contraception
* Presence of ferromagnetic material in the cranium except in the mouth, including metal fragments from occupational exposure, and surgical clips in or near the brain
* Cardiac or neural pacemakers or implanted medication pumps
* Receptive aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Baseline, Immediately post-intervention
  This is a quantitative measure of motor recovery, coordination, and speed.

SECONDARY OUTCOMES:
Action Research Arm Test | Baseline, Immediately post-intervention
  This test measures changes in the upper extremity and consists of four specific tests to measure grasp, grip, pinch, and gross movement.
Stroke Impact Scale | Baseline, Immediately post-intervention
  This is a self-report that assesses strength, hand function, activities of daily living, mobility, communication, emotion, memory and thinking, and participation.
Cortical motor map volume | Baseline, Immediately post-intervention
  This is performed using non-invasive transcranial magnetic stimulation to determine which parts of the brain control a muscle in the arm or hand.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky at Cardinal Hill Rehabilitation Hospital, Lexington, Kentucky, United States